CLINICAL TRIAL: NCT00173017
Title: The Physiological Impact of N95 Masks on Medical Staff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 9261700712
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-06

CONDITIONS: Hypoxemia; Hypercapnia
Keywords: N95 mask; medical staff; hypoxemia; hypercapnia; neurological study
MeSH Terms: conditions — Hypoxia; Hypercapnia

INTERVENTIONS:
Device: wearing N95 masks

SUMMARY:
Wearing N95 masks may have adverse physical effect on medical staff

DETAILED DESCRIPTION:
Wearing N95 masks results in hypooxygenemia and hypercapnia which reduce working efficiency and the ability to make correct decision.

Medical staff are at increased risk of getting 'Severe acute respiratory syndrome'(SARS), and wearing N95 masks is highly recommended by experts worldwide. However, dizziness, headache, and short of breath are commonly experienced by the medical staff wearing N95 masks. The ability to make correct decision may be hampered, too. The purpose of the study was therefore to evaluate the physiological impact of N95 mask on medical staff.

ELIGIBILITY:
Inclusion Criteria:

* medical staff

Exclusion Criteria:

* pregnancy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2003-08; Study Completion 2005-06

PRIMARY OUTCOMES:
EEG change, ABG change, change in scores of attention test, etc

SECONDARY OUTCOMES:
symptoms wearing N95 masks

CONTACTS AND LOCATIONS:
Overall Officials: Tze-Wah Kao, master, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan